CLINICAL TRIAL: NCT00397709
Title: Short-Course Isoniazid and Rifampin Compared With Isoniazid for Latent Tuberculosis Infection: A Randomized Clinical Trial.
Brief Title: Short-Course Isoniazid and Rifampin Compared With Isoniazid for Latent Tuberculosis Infection
Status: Terminated | Phase: Phase 4 | Type: Interventional
Sponsor: Hospital Virgen de la Luz (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TBQXCU2; TBQXPNCU1
Record Dates: First submitted 2006-11-07; First posted 2006-11-09 (Estimated); Last update posted 2008-12-31 (Estimated); Status verified 2006-11

CONDITIONS: Tuberculosis
Keywords: Latent tuberculosis infection.; Isoniazid.; Rifampin.; Clinical trial.; treatment of latent tuberculosis infection
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis | interventions — Isoniazid; Rifampin

INTERVENTIONS:
Drug: I ( isoniazid), II (isoniazid + rifampin )

SUMMARY:
The objective of the study was to compare the compliance and the side effects of a short course to treatment of latent tuberculosis infection during 3 months(isoniazid plus rifampin)group I, with the standard course for 6 months(isoniazid)group II .Prospective, comparative, randomized and open trial of patients with positive TST and the suitable criteria for treatment, in accordance with the guidelines of the CDC, excluding HIV infection. 105 patients were included. In Conclusion, a short course with isoniazid plus rifampin during 3 months shown better compliance with a lower percentage of abandonment that the course 6H. Tolerance is similar in the two courses.

DETAILED DESCRIPTION:
Introduction: The objective of the study was to compare the compliance and the side effects of a short course to treatment of latent tuberculosis infection during 3 months with the standard course for 6 months.

Methods: Prospective, comparative, randomized and open trial of patients with positive TST and the suitable criteria for treatment, in accordance with the guidelines of the CDC, excluding HIV infection. the group I was assigned to isoniazid (H) at a dose of 300 mg per day for 6 months and the group II was assigned to isoniazid at a dose of 300 mg per day plus rifampin (R) (600 mg per day) for 3 months. The patients were followed for five years.

Results: 105 patients were included, of which 9 refused the treatment; 45 patients were included in the group I and 51 patients in the group II. Both groups were comparable at base level. The hepatotoxicity was 44% in the group 6H and 29% in the group 3HR (p = 0,07). The hepatotoxicity was severe in 6.7% in the group 6H and 5.8% in the group 3HR; these obliged the suspension of treatment in 4.4% and 1.9%, respectively (p =NS). The proportion of patients who completed the study treatment was 75.6% of the patients in the group 6H, and 90.2% in the group 3HR (p = 0,05). Only a case of tuberculosis was detected in the second month treatment with 6H.

Conclusion: In the treatment of latent tuberculosis infection, a short course with isoniazid plus rifampin during 3 months shown better compliance with a lower percentage of abandonment that the course 6H. Tolerance is similar in the two courses.

ELIGIBILITY:
Inclusion Criteria:

* patients with positive TST and the suitable criteria for treatment, in accordance with the guidelines of the CDC:

Exclusion Criteria:

* HIV infection.
* Hepatopathy
* Previous treatment of of latent tuberculosis infection.
* Allergy to drugs.

Ages: 16 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 228
Dates: Start 1996-03; Study Completion 2006-02

PRIMARY OUTCOMES:
to compare the compliance
to compare the side effects

SECONDARY OUTCOMES:
Development of tuberculosis

CONTACTS AND LOCATIONS:
Overall Officials: Maria Paloma Geijo Martinez, MD, Principal Investigator — Unidad MI-Infecciosas. Hospital Virgen de la Luz. Cuenca 16002 Spain
Locations (1):
- Maria Paloma Geijo Martinez. Hospital Virgen de la Luz, Cuenca, Cuenca, Spain

REFERENCES:
- [Derived] Geijo MP, Herranz CR, Vano D, Garcia AJ, Garcia M, Dimas JF. [Short-course isoniazid and rifampin compared with isoniazid for latent tuberculosis infection: a randomized clinical trial]. Enferm Infecc Microbiol Clin. 2007 May;25(5):300-4. doi: 10.1157/13102264. Spanish. PMID 17504682
- See also: Page of infectious diseases of the region with studies on TB — http://sescam.jccm.es/web1/home.do